CLINICAL TRIAL: NCT04363866
Title: A Randomized-Control Pilot Study to Assess Hydroxychloroquine in Patients Infected With SARS-CoV-2 (COVID-19)
Brief Title: Assessing Hydroxychloroquine in Patients With SARS-CoV-2 (COVID-19)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: discontinued in favor of more promising directions that may benefit patients
Sponsor: Oregon Health and Science University (Other)
Collaborators: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Marcel Curlin, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00021303
Record Dates: First submitted 2020-04-24; First posted 2020-04-27 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: SARS-CoV-2; COVID-19; Hydroxychloroquine; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded Study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Experimental): 400 mg bid (PO) Day 1, followed by 200 mg bid (PO) Day 2 through Day 5
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Placebo pill bid (PO) Day 1 through Day 5 of the treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine is more polar, less lipophilic, and has more difficulty diffusing across cell membranes than the parent compound, chloroquine. These characteristics result in hydroxychloroquine having a longer half-life, comparatively lower toxicity to chloroquine, as well as fewer concerns pertaining to drug-drug interactions
  Arms: Hydroxychloroquine
Drug: Placebo — A placebo is a pill that looks like the study drug but has no real medicine in it.
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blinded, placebo-controlled, pilot study to assess the preliminary efficacy and safety of hydroxychloroquine for the treatment of patients with lower respiratory tract SARS-CoV-2 infection.

DETAILED DESCRIPTION:
A total of 40 participants are planned for enrollment. Those enrolled into this study will be randomized 1:1 to receive either hydroxychloroquine or placebo control.

Participants will receive their study intervention for 5 days, after which they will be considered off protocol- directed therapy and receive medical management of their disease according to institutional standards. Participants may be followed for up to 180 days from initiating protocol therapy for clinical outcome, after which they will discontinue study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document.
2. Individuals aged ≥ 18 years of all races and ethnic groups.
3. Must have documented positive test result for SARS-CoV-2 (COVID19), or high clinical suspicion for SARS-CoV-2 based on presence of typical clinical findings (e.g., fever, respiratory symptoms, pulmonary abnormalities on chest X-ray or CT scan), lack of alternative diagnosis, and history of exposure to a known case of SARS-CoV- 2 infection within the past 14 days
4. Not receiving institutional therapy for treatment of SARS-CoV-2, including (but not limited to) remdesivir, chloroquine, hydroxychloroquine, or any other investigational agent(s).
5. Must meet at least one of the following clinical stratifications:

   1. Have at least 1 minor criterion per ATS criteria (refer to Appendix A), or
   2. Have fever, respiratory symptoms, with pneumonia visible on chest imaging (e.g., X-ray or computed tomography [CT]), or
   3. High risk for poor outcome, as defined by any one of the following:

   i. Age ≥ 60 years old ii. Underlying medical comorbidities, defined as:
   * Serious cardiovascular disease
   * Poorly controlled diabetes (i.e., A1c levels >7%)
   * Chronic kidney disease requiring dialysis
   * Significant liver disease (Pugh-Child B or C)
   * Severe obesity (body mass index [BMI] ≥ 40)
   * Chronic respiratory disease (e.g., COPD)
   * Hypertension, defined as blood pressure ≥ 140 / 90 mmHg iii. Solid organ or stem cell transplant recipient iv. Diagnosis of solid or hematologic malignancy being treated with systemic chemotherapy v. Receipt of biologic agent or prednisone > 0.5 mg/kg/day (or equivalent)
6. Patient must be within 5 days of symptom onset, as determined by clinical team.
7. Participants with preexisting auditory damage are allowed.
8. Participants with a history of epilepsy are allowed.
9. Female participants of childbearing potential (FOCBP) must have a negative serum or urine pregnancy test (per institutional standards) prior to the start of study drug.
10. FOCBP must agree to use highly-effective method(s) of contraception (Appendix B) during the study and for 1 months after the last dose of study drug. FOCBP are those who have not been surgically sterilized or have not been free from menses for >1 year without an alternative medical cause.
11. Male participants must agree to use an adequate method of contraception (Appendix B) starting with the first dose of study therapy through at least 1 months after the last dose of study drug.
12. Participant must agree to not breastfeed during the study or for 30 days after the last dose of study treatment.

Exclusion Criteria:

1. The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study.
2. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
3. Psychiatric illness/social situations, or any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of participant safety or study results, or substantially increase risk of incurring AEs, or compromise the ability of the patient to give written informed consent.
4. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or participants with congenital long QT syndrome
5. Patients with Myesthenia Gravis or other neuromuscular disorders
6. Patients with history of psoriasis.

   a. May be waived at the discretion of the PI
7. Patients with history of porphyria

   a. May be waived at the discretion of the PI
8. Concomitant use of other antiviral agents for the study's duration, but may be waived at discretion of the Principal Investigator
9. Hypersensitivity to the study agent, or any of its excipients.
10. Females who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Clinical Status at Day 5 Assessed by a 6-Point Ordinal Scale | Day 5
  A 6-point ordinal scale ranging from "Death" to "Not hospitalized with full resumption of normal activities" is used to evaluate differences in the clinical status between participants that receive placebo vs hydroxychloroquine

SECONDARY OUTCOMES:
Number of Participants with Detectable SARS-CoV-2 Virus from Day 0 to Day 28 and at Day 5 | Day 0 to Day 28 and at Day 5
  Assess differences in SARS-CoV-2 viral shedding between participants that receive placebo vs hydroxychloroquine
Toxicity of Study Drug Assessed by Incidence of Adverse Events | Day 0 to Day 28
  Assess by incidence of Grade 3, Grade 4, and Serious Adverse Events (AEs)

OTHER OUTCOMES:
Duration of Initial Hospitalization | Day 0 to Day 28
  Assess length of hospitalization
Mortality During Follow-Up | Day 0 to Day 28
  Assess number of deaths during study follow-up
Mortality During Initial Hospitalization | Day 0 to Day 28
  Assess number of deaths in the hospital during initial hospitalization
Incidence of New Hospital Resource Utilization | Day 0 to Day 28
  Assessing utilization of hospital resources
Duration of Hospital Resource Utilization | Day 0 to Day 28
  Assessing duration of hospital resource utilization
Changes in Cytokine Profile | Day 0 to Day 28
  Provide preliminary characterization of differences in inflammatory response between participants that receive placebo vs hydroxychloroquine

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Curlin, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after the identification
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Anyone who wishes to access the data for any purpose. Data may be obtained by contacting the corresponding author of the relevant publication